CLINICAL TRIAL: NCT00280085
Title: Pancreatic Beta-Cell Mass And Function Quantification By Means Of Perfusion Imaging
Brief Title: The Aim is to Estimate the Total Amount of Insulin-producing Cells in the Pancreas by MRI.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Explanation provided in detailed descriptiong section of record.
Sponsor: Pfizer (Industry)
Collaborators: Yale University (Other)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A9001280
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2008-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Magnetic Resonance Spectroscopy; Glucose Clamp Technique; Arginine

INTERVENTIONS:
Procedure: MR imaging
Procedure: Glucose clamp
Drug: Arginine
  Other Names: R-Gene 10

SUMMARY:
Assess pancreatic beta cell function using MR imaging.

DETAILED DESCRIPTION:
The study was terminated on July 31st, 2007. The study was discontinued, as we have not met the primary end point, differentiation between normal volunteers and subjects with type 1 diabetes mellitus. There were no safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Normal Volunteers
* T1DM and T2DM subjects

Exclusion Criteria:

* Concomitant severe conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-12; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pancreatic perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Hirshberg B, Qiu M, Cali AM, Sherwin R, Constable T, Calle RA, Tal MG. Pancreatic perfusion of healthy individuals and type 1 diabetic patients as assessed by magnetic resonance perfusion imaging. Diabetologia. 2009 Aug;52(8):1561-5. doi: 10.1007/s00125-009-1406-8. Epub 2009 Jun 3. PMID 19488737
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001280&StudyName=The%20aim%20is%20to%20estimate%20the%20total%20amount%20of%20insulin-producing%20cells%20in%20the%20pancreas%20by%20MRI.